CLINICAL TRIAL: NCT05518370
Title: The Effect of Hippotherapy Simulator on Sitting Balance, Trunk Control and Upper Extremity Skills in Cerebral Palsy
Brief Title: The Effect of Hippotherapy Simulator in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Demet GÖZAÇAN KARABULUT, Assistant Professor, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIBTU-FTR-DGK-1
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Hippotherapy simulator
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hippotherapy simulator training group (Experimental): Hippotherapy simulator training group will receive a traditional physiotherapy and hippotherapy simulator training, two days a week for a total of 8 weeks (30 minutes traditional physiotherapy session+15 minutes hippotherapy simulator training).
  Interventions: Other: Hippotherapy simulator training; Other: Traditional physiotherapy
- Traditional physiotherapy group (Active Comparator): Traditional physiotherapy group individuals will be given a traditional physiotherapy two days per week for a total of 8 weeks (traditional physiotherapy session will last 45 minutes).
  Interventions: Other: Traditional physiotherapy

INTERVENTIONS:
Other: Hippotherapy simulator training — Hippotherapy simulator training will be designed for the individual basis.
  Arms: Hippotherapy simulator training group
Other: Traditional physiotherapy — Traditional physiotherapy within a specific program

SUMMARY:
Hippotherapy simulators imitate the passive movements of the horse, producing simple movements similar to those of the horse. Hippotherapy simulators are intended to improve sitting balance, postural control and trunk balance.

The aim of this study was to research the therapeutic effects of hippotherapy simulator on sitting balance, trunk control and upper extremity skills in individuals with Cerebral Palsy (CP).

DETAILED DESCRIPTION:
Spastic CP will be participate the study between the ages of 4 and 18 years. Children's classified with GMFCS and MACS.

The eligible participants will be allocated two groups, including hippotherapy simulator training group and traditional physiotherapy control group. All the assessments will be performed before and after the training in the 8-week training groups.

The control group individuals will be given a traditional physiotherapy two days per week for a total of 8 weeks (traditional physiotherapy session will last 45 minutes). Hippotherapy simulator training group will receive a traditional physiotherapy and hippotherapy simulator training, two days a week for a total of 8 weeks (30 minutes traditional physiotherapy session+15 minutes hippotherapy simulator training). All sessions will be performed in the clinic with the specialist physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Spastic Cerebral Palsy voluntary participation
* Age between 4-18 years,
* GMFCS Level I-II-III
* MACS Level I-II-III
* Have the ability to sit upright with support

Exclusion Criteria:

* Not voluntary to participate in the research,
* Botox in the last 6 months
* Hip or spine surgeries in the last 6 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | At Baseline
  Assessing functional level and motor function. Gross motor functions of children with CP are classified in five levels with GMFCS. This is a classification system based on the child's self-initiated movements with emphasis on sitting, displacement and mobility.
Manuel ability classification system (MACS) | At Baseline
  This is a classification system based on the grasping and releasing objects in daily life, and how they use their hands while holding objects. It is classify the hand skills of children with CP between the ages of 4-18.Children with CP are classified in five levels with MACS. The higher level indicates worse hand function
Change from Baseline Gross Motor Function Measure-88 at 8 weeks | Change from Baseline at 8 weeks
  It is used to show gross motor functions and changes in these functions. It consists of five main sections. Each section can be used by calculating separately within itself. The total score ranges from 0 to 100, with a high score indicating better function.
Change from Baseline Trunk Control Measurement Scale at 8 weeks | Change from Baseline at 8 weeks
  This scale consists of two main parts as dynamic and static sitting balance. The scale consists of 15 questions. The scoring of the items is 0, 1, 2 or 3. The total score ranges from 0 to 58, with a high score indicating better trunk control.
Change from Baseline Pediatric Evaluation of Disability Inventory at 8 weeks | Change from Baseline at 8 weeks
  The Pediatric Evaluation of Disability Inventory (PEDI) is designed for the functional evaluation of children with special needs. This will be used to evaluate functional ability and performance. 0: can not do, 1: can do in the form of scoring is done. At the end of the evaluation, the points of the related section are collected. Higher score indicates a better level of functional independence.
Change from Baseline ABILHAND-Kids at 8 weeks | Change from Baseline at 8 weeks
  Abilhand Kids evaluates manual ability in children with upper extremity disorders. It consists of 21 items and confirmed in CP. The lowest score that can be obtained from the scale is 21 and the highest score is 63. It can be stated that higher scores correspond to more difficulty in activities.
Change from Baseline The Jebsen Taylor Hand Function Test at 8 weeks | Change from Baseline at 8 weeks
  The Jebsen Taylor Hand Function Test (JTHFT) will be used to evaluate hand function in daily life. Both hands are tested separately. The time for all activities is recorded with a stopwatch. Higher duration indicates worse hand function.

CONTACTS AND LOCATIONS:
Overall Officials: Demet GÖZAÇAN KARABULUT, Study Director — Gaziantep Islam Science and Technology University
Locations (1):
- Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gozacan Karabulut D, Numanoglu Akbas A. The effect of horse riding simulator on upper extremity skills, trunk control and functionality in cerebral palsy: a randomized controlled trial. Disabil Rehabil. 2025 Apr;47(7):1725-1732. doi: 10.1080/09638288.2024.2380785. Epub 2024 Jul 18. PMID 39022889